CLINICAL TRIAL: NCT00856089
Title: Prevalence of Methicillin-resistant Staphylococcus Aureus (MRSA) in a Medical Center and Efficacy of Altabax in Clearing MRSA Nasal Colonization
Brief Title: Efficacy Study of Altabax to Clear Methicillin-resistant Staphylococcus Aureus (MRSA) Nasal Colonization
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study is withdrawn and no one enrolled due to changes in personnel
Sponsor: Ochsner Health System (Other)
Collaborators: Tulane University School of Medicine (Other); GlaxoSmithKline (Industry)
Responsible Party: Russell W Steele, MD, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT112759
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
MeSH Terms: interventions — retapamulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Retapamulin (Experimental)
  Interventions: Drug: Retapamulin

INTERVENTIONS:
Drug: Retapamulin — Retapamulin ointment, 1%, apply a thin layer, BID for 5 days
  Other Names: Altabax

SUMMARY:
The purpose of the study is to determine whether Altabax (retapamulin ointment, 1%) is effective in the treatment of methicillin-resistant Staphylococcus aureus (MRSA) nasal colonization. The hypothesis is that the prevalence of MRSA increases as a function of increasing clinical exposure and that the topical antibiotic Altabax is efficacious in clearing MRSA nasal colonization. The prevalence of MRSA nasal colonization among Tulane University medical students and residents and physicians of Tulane Medical Center and Ochsner Medical Center will be investigated. A total of 300 subjects will be recruited for the study. After giving informed consent, subjects will be swabbed to obtain specimens for culture and asked to complete a short survey to assess risk factors. Swabs will be used to directly inoculate three types of plates: CHROMagar MRSA plates, Spectra MRSA plates, and TSA with sheep blood plates. After appropriate incubation, Staph latex slide tests will be done and then results confirmed with cefoxitin disk susceptibility testing. MRSA positive subjects will be offered a treatment protocol with the topical antibiotic Altabax (retapamulin ointment, 1%) to be applied as a thin layer to the anterior nares twice daily for 5 days. After the 5-day treatment is complete, subjects will be retested for the presence of MRSA at day 7, day 12, day 30, and day 90. For this portion of the study, all cultures will additionally undergo disk susceptibility testing for retapamulin, erythromycin, clindamycin (including D-test), trimethoprim sulfa, and mupirocin (5 mcg and 20 mcg disks). In addition, Etests for retapamulin and mupirocin will be done. Genetic isolates will be characterized by rep-PCR pre-treatment and post-treatment. Data will be analyzed for MRSA prevalence and risk factor associations with MRSA colonization. Of those subjects found to be MRSA positive, data from the follow-up cultures will be used to assess the efficacy of Altabax in clearing MRSA nasal colonization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be either a student, resident, or physician at Tulane University or be a resident or physician at Ochsner Medical Center.

Exclusion Criteria:

* Subjects who are pregnant or who are presently taking antibiotics or require treatment with systemic antibiotics at anytime during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Eradication of MRSA nasal colonization | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Russell W Steele, MD, Principal Investigator — Ochsner Health System
Locations (2):
- United States (2):
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana